CLINICAL TRIAL: NCT03407768
Title: Role of Individualized Intervention(s) on Quality of Life and Adherence to Adjuvant Endocrine Therapy in Premenopausal Women With Early-Stage Breast Cancer
Brief Title: Role of Individualized Intervention(s) in Hormone-Receptor Positive Early-stage Breast Cancer
Acronym: MyCHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Shahid Ahmed, MD, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 348455
Record Dates: First submitted 2017-10-24; First posted 2018-01-23 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Premenopausal Breast Cancer; Hormone Receptor Positive Tumor
Keywords: Premenopausal breast cancer; Individualized interventions; Exercise; Combination hormone therapy; Massage therapy; Yoga; Acupuncture; Treatment tolerance; Treatment adherence; Adverse effects; Quality of life
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized interventions (Other): Exercise, Yoga, massage therapy, acupuncture, and others
  Interventions: Behavioral: Individualized interventions

INTERVENTIONS:
Behavioral: Individualized interventions — A participant will be able to select one or more (or no intervention) based on her preferences.
  Individualized exercise program Yoga and mindfulness Massage therapy Acupuncture Others: Women who are not interested in any above intervention but like to explore other interventions will be offered material pertinent to their choice of complimentary techniques.

SUMMARY:
Although combination endocrine therapy has been associated with significant reduction in risk of recurrence in younger women with hormone receptor positive breast cancer, it has been associated with more adverse effects and decline in quality of life (QOL). Various behavioral and complementary interventions can be effective in reducing treatment-related side effects. The study aims to evaluate if individually-tailored behavioral and complementary interventions could improve treatment tolerance and adherence in women with early stage breast cancer. This benefit will be assessed primarily by change in QOL and secondarily by adherence to adjuvant endocrine treatment.

DETAILED DESCRIPTION:
Recent evidence suggest that ovarian suppression in combination with exemestane compared with tamoxifen alone has been associated with significant reduction in risk of breast cancer recurrence in premenopausal women with high risk estrogen or progesterone receptor positive breast cancer. However, combination therapy has been associated with more adverse effects, poor treatment adherence, and decline in quality of life (QOL). Various behavioral and complementary interventions such as exercise, yoga, acupuncture, and massage therapy can be effective to reduce treatment-related side effects and thereby to improve QOL. Nevertheless, there is a paucity of evidence about effect of individualized behavioral and complementary interventions in younger women who are treated with combination endocrine therapy. The study aims to evaluate if younger women with early stage breast cancer treated with combination endocrine therapy could benefit from individualized behavioral and complementary intervention (s) during their treatment. This benefit will be assessed primarily by change in QoL and cognitive function from the baseline measurement and secondarily by adherence to adjuvant endocrine treatment. Furthermore, the study will explore correlation between selection of intervention(s) and various socio-demographic and clinical factors. Forty premenopausal women with early stage breast cancer treated with combination endocrine therapy will be recruited over a two year period in Saskatchewan with a median follow up period of about two years. All participants will be provided a list of interventions that alone or in combination could be helpful to improve treatment tolerance to hormonal therapy. A participant will be able to select one or more intervention based on her preferences. The QOL and cognitive function will be assessed every three months using Functional Assessment of Cancer Therapy - Breast Symptom Index (FACT-B), FACT - Endocrine System (FACT-ES), and FACT-Cognitive Function scales. Treatment adherence will be monitored monthly basis. Individually-tailored behavioral and complementary interventions could promote self-management and empower the women with early stage breast cancer to manage treatment related side effects.

ELIGIBILITY:
Inclusion Criteria:

• Premenopausal women with histologically-proven, completely resected, hormone receptor-positive (defined as ER≥10% and/or PgR≥10%) stage 1, 2, and 3 invasive breast cancer who are treated with combination of anti-estrogen therapy (LHRH agonist and an aromatase inhibitor or tamoxifen)

Exclusion Criteria:

* Post-menopausal women
* Women who are on single agent endocrine therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - Breast Symptom Index (FACT-B) | Up to three years from the time of enrolment
  For global assessment of quality of life of women with breast cancer

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - Endocrine System (FACT-ES) | Up to three years from the time of enrolment
  For the assessment of quality of life of women with breast cancer on endocrine therapy
Functional Assessment of Cancer Therapy - (FACT)-Cognitive | Up to three years from time of enrolment
  For the assessment of self-reported cognitive function
Treatment discontinuation rate | Up to three years from the time of enrolment
  Rate of combination of endocrine treatment at 3 year.

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Ahmed, MD, PhD, Principal Investigator — University of Saskatchewan
Locations (2):
- Canada (2):
  - Allan Blair Cancer Center, Regina, Saskatchewan
  - Saskatoon Cancer Center, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No
If requested in future after meeting all the regulatory requirement data will be shared.